CLINICAL TRIAL: NCT06044298
Title: The Impact of Frailty on Adverse Events in Patients Undergoing Gastrointestinal Procedural Sedation: a Multicentre, Prospective, Observational Study(FRAEPS Study)
Brief Title: Advers Events in Patients Undergoing Gastrointestinal Procedural Sedation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Cansabuncu, Medical Doctor, Uludag University
Other Study IDs: 2023-16/23
Record Dates: First submitted 2023-08-22; First posted 2023-09-21 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Sedation Complication; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastrointestinal procedural sedation: Investigators will include in our study patients aged 60 and over who have been evaluated in the pre-anesthesia clinic for procedures such as endoscopy, colonoscopy, ERCP, PEG, EUS, and ESD, and who have received sedation by an anesthesiologist. Patients will be assessed for frailty prior to the procedure; during and after the procedure, respiratory monitoring (SpO2, capnography) will be closely observed, and they will be contacted by phone three days later.
  Interventions: Other: procedural sedation

INTERVENTIONS:
Other: procedural sedation — "Participants, adverse events during and after gastrointestinal procedures with sedation administered were observed and recorded. No intervention was performed."

SUMMARY:
Investigators will include in our study patients aged 60 and over who have been evaluated in the pre-anesthesia clinic for procedures such as endoscopy, colonoscopy, ERCP, PEG, EUS, and ESD, and who have received sedation by an anesthesiologist. Patients will be assessed for frailty prior to the procedure; during and after the procedure, respiratory monitoring (SpO2, capnography) will be closely observed, and they will be contacted by phone three days later.

Primary goal of the study is to prospectively investigate the incidence of peri-procedural complications (desaturation, bradycardia, hypotension, etc.) in elderly patients undergoing gastrointestinal procedural sedation, and to assess its relationship with detected frailty using the FRAIL scale.Secondary goals of the study are to identify risk factors for adverse events, examine the relationship of these factors with 'ASA score - age and frailty scale', and determine their impact on the incidence of adverse events. Additionally, investigators aim to research the effects of capnography-based respiratory monitoring on adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older patients
* ASA physical state I -IV
* Patients who are qualified to give written informed consent
* Elective gastrointestinal interventions performed under the care of the anesthesia team (such as gastroscopy, colonoscopy).

Exclusion Criteria:

* ASA IV patients
* Patients using sedative agents / Patients already sedated for other purposes
* Non-consenting patients
* Patients with any upper airway obstructive pathology or a history of difficult airway
* Emergency procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — over 60 years old
Study Population: Investigators intend to include in the study patients aged 60 and above who have been evaluated in the pre-anesthesia clinic prior to procedures (such as endoscopy, colonoscopy, ERCP, PEG, EUS, ESD) and have received sedation by an anesthesiologist.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Advers event,fraility | first day
  The primary aim of the FRAEPS study is to prospectively investigate the incidence of peri-procedural complications in elderly patients undergoing gastrointestinal procedural sedation, as well as the relationship between these complications and the frailty assessed by the FRAIL (Fatigue, Resistance, Ambulation, Illness, Loss of weight) scale. FRAIL Scale is rated from 0-5. (Non frail:0, prefrail:1-2, frail: 3-5)

SECONDARY OUTCOMES:
Precedural advers event | First day
  The secondary objectives of the FRAEPS study are to determine risk factors for adverse events, explore the relationship between ASA (American Society of Anesthesiologist) classification and frailty scale.
Capnography and side effects | First day
  Investigators intend to investigate the effects of monitoring respiratory activity through capnography on the improvement of procedural side effects.
Postprocedural advers event | Third day
  In the early post-procedural period (Day 3), investigators will assess whether the patient has returned to their pre-procedure state, whether they require additional support, and determine rates of readmission.

CONTACTS AND LOCATIONS:
Overall Officials: suna gören, Principal Investigator — Uludag University
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)